COMIRB APPROVED For Use 16-Jul-2021

**Principal Investigator: Matthew Haemer MD MPH** 

COMIRB No: 21-3712 Version Date: 7.16.2021

Study Title: Family Inclusive Childhood Obesity Treatment Designed for Low Income and Hispanic Families

You are being asked to be in a research study. This form provides you with information about the study. A member of the research team will describe this study to you and answer all of your questions. Please read the information below and ask questions about anything you don't understand before deciding whether or not to take part.

### Why is this study being done?

This study is designed to learn more about program delivery costs.

You are being asked to be in this research study because you are staff (health educator or fitness trainer) delivering the Healthy Living Program (HeLP) at a Rec Center or delivery site.

Up to 20 HeLP staff will participate in the study.

# What happens if I join this study?

If you join the study, team members will observe the time it takes for you to complete 3 entire HeLP sessions and individual portions of the program.

Study participation will last up to 4 years.

#### What are the possible discomforts or risks?

Discomforts you may experience while in this study include feeling uncomfortable being observed by research staff.

#### What are the possible benefits of the study?

This study is designed for the researcher to learn more about the cost of delivering the Healthy Living Program. This study is not designed to benefit you directly.

# Who is paying for this study?

This research is being paid for by the *National Institutes of Health (NIH)*.

### Will I be paid for being in the study? Will I have to pay for anything?

You will not be paid to be in the study. Consent Template Social and Behavioral CF-156, Effective 10-24-18 Page **1** of **3** 

#### **Consent Form**

It will not cost you anything to be in the study.

# Is my participation voluntary?

Taking part in this study is voluntary. You have the right to choose not to take part in this study. If you choose to take part, you have the right to stop at any time. If you refuse or decide to withdraw later, you will not lose any benefits or rights to which you are entitled.

### Who do I call if I have questions?

The researcher carrying out this study is Dr. Matthew Haemer. You may ask any questions you have now. If you have questions later, you may call Dr. Matthew Haemer at 720-777-7474 or Program Manager Emily Steen at 303-214-8091.

You may have questions about your rights as someone in this study. You can call Dr. Matthew Haemer with questions. You can also call the Multiple Institutional Review Board (IRB). You can call them at 303-724-1055.

# **Certificate of Confidentiality**

This study has been issued a Certificate of Confidentiality from the federal government to help protect your privacy. The Certificate prohibits the researchers from disclosing your name, or any identifiable information, document or biospecimen from the research, with the exceptions listed below. A certificate provides protections against disclosing research information in federal, state, or local civil, criminal, administrative, legislative or other proceedings.

These protections apply only to your research records. The protections do not apply to your medical records.

The researchers may disclose your name or identifiable information, document or biospecimen, under the following circumstances:

- To those connected with the research,
- If required by Federal, State or local laws,
- If necessary for your medical treatment, with your consent,
- For other scientific research conducted in compliance with Federal regulations,
- To comply with mandated reporting, such as a possible threat to harm yourself or others, reports of child abuse, and required communicable disease reporting, or
- Under other circumstances with your consent.

#### **Consent Form**

A Certificate of Confidentiality does not protect information you or a member of your family voluntarily release.

# Who will see my research information?

We will do everything we can to keep your records a secret. It cannot be guaranteed.

Both the records that identify you and the consent form signed by you may be looked at by others.

- Federal agencies that monitor human subject research
- Human Subject Research Committee
- The group doing the study
- The group paying for the study
- Regulatory officials from the institution where the research is being conducted who want to make sure the research is safe

The data we collect will be used for this study but may also be important for future research. Your data may be used for future research or distributed to other researchers for future study without additional consent if information that identifies you is removed from the data.

The results from the research may be shared at a meeting. The results from the research may be in published articles. Your name will be kept private when information is presented.

### Agreement to be in this study

I have read this paper about the study or it was read to me. I understand the possible risks and benefits of this study. I know that being in this study is voluntary. I choose to be in this study: I will get a copy of this consent form.

| Signature: | Date: |
|----------------------------|-------|
| Print Name: | |
| Consent form explained by: | Date: |
| Print Name: | |